CLINICAL TRIAL: NCT00358046
Title: A Phase 2, Randomized, Dose-Ranging, Single-Blind, Efficacy and Tolerability Study of ILY101 in Patients With Chronic Kidney Disease With Hyperphosphatemia on Hemodialysis
Brief Title: Efficacy and Tolerability of ILY101 in Dialysis Patients With Hyperphosphatemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ilypsa (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILY-1201
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Kidney Diseases; Renal Insufficiency
Keywords: Hyperphosphatemia; Chronic kidney disease; Dialysis; Hyperphosphatemia in CKD patients on dialysis
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Hyperphosphatemia; Renal Insufficiency, Chronic

INTERVENTIONS:
Drug: ILY101

SUMMARY:
This is a randomized, dose-ranging, efficacy and tolerability study in chronic kidney disease patients with hyperphosphatemia on hemodialysis. Patient participation in the study is approximately 10 weeks in duration.

DETAILED DESCRIPTION:
Hyperphosphatemia is associated with abnormally high blood concentrations of phosphorus. Normally, phosphorus in the body is excreted into urine via the kidneys, but this process is impaired when renal function is reduced. Hyperphosphatemia occurs in many patients with renal insufficiency, especially those on dialysis. High blood phosphorus concentrations trigger various complications caused by phosphorous interaction with blood calcium or parathyroid hormones, and makes patients more prone to calcium deposition in soft tissues such as the coronary arteries, increasing the risk of ischemic heart disease. ILY101 is a non-absorbed, metal-free polymer that binds phosphorus in the gastrointestinal tract, allowing for excretion of phosphorus. It is therefore anticipated to ameliorate hyperphosphatemia by reducing the absorption of phosphorus from the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients on dialysis
* Prior successful use of phosphate binder
* Signed informed consent

Exclusion Criteria:

* Previous intolerance to polymer-based phosphate binders
* Kidney transplant planned within 3 months
* Pregnant or lactating women, or women of child bearing potential not using an acceptable form of birth control
* Clinically significant liver disease
* History of bowel obstruction or other significant gastrointestinal disorder

Additional study entry criteria will be evaluated during initial screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Guido Smeets, MD, Study Director — Ilypsa
Locations (18):
- United States (18):
  - Clinical Study Site, Mobile, Alabama
  - Clinical Study Site, Mountain View, California
  - Clinical Study Site, Riverside, California
  - Clinical Study Site, San Diego, California
  - Clinical Study Site, Thornton, Colorado
  - Clinical Study Site, Ocala, Florida
  - Clinical Study Site, Palm Beach Gardens, Florida
  - Clinical Study Site, Pembroke Pines, Florida
  - Clinical Study Site, Des Moines, Iowa
  - Clinical Study Site, Baton Rouge, Louisiana
  - Clinical Study Site, Rochester, New York
  - Clinical Study Site, Allentown, Pennsylvania
  - Clinical Study Site, Houston, Texas
  - Clinical Study Site, San Antonio, Texas
  - Clinical Study Site, Provo, Utah
  - Clinical Study Site, Salt Lake City, Utah
  - Clinical Study Site, Norfolk, Virginia
  - Clinical Study Site, Appleton, Wisconsin

REFERENCES:
- See also: Related Info — http://www.ilypsa.com